CLINICAL TRIAL: NCT00806598
Title: Phase II Study of Combination of Thymoglobulin, Cyclosporine, Methylprednisone, and Granulocyte Colony-stimulating Factor (GCSF) in Patients With Newly Diagnosed Aplastic Anemia or With Hypoplastic or Low/Intermediate-1 Risk Myelodysplastic Syndrome
Brief Title: Thymoglobulin and Cyclosporine in Patients With Aplastic Anemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0115
Record Dates: First submitted 2008-12-09; First posted 2008-12-11 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Myelodysplastic Syndrome; Aplastic Anemia
Keywords: Myelodysplastic Syndrome; Aplastic Anemia; Thymoglobulin; Cyclosporine; Methylprednisolone; G-CSF
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Aplastic | interventions — thymoglobulin; Antilymphocyte Serum; Cyclosporine; Methylprednisolone; Methylprednisolone Hemisuccinate; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thymoglobulin + Cyclosporin (Experimental): Combination of Thymoglobulin 3.5 or 2.5 mg/kg/day intravenous (IV) for 5 days + Methylprednisone 1 mg/kg/day IV for 5 days, before each dose Thymoglobulin + Cyclosporin 5 mg/kg orally for 6 months following Thymoglobulin + Granulocyte - Colony Stimulating Factor (G-CSF) 5 microgram/kg subcutaneously daily up to 3 months
  Interventions: Drug: Thymoglobulin; Drug: Cyclosporine; Drug: Methylprednisolone; Drug: G-CSF

INTERVENTIONS:
Drug: Thymoglobulin — 3.5 or 2.5 mg/kg/day IV for 5 days
  * Aplastic anemia patients receive 3.5 mg/kg/day for 5 days
  * MDS patients <55 years receive 3.5 mg/kg/day for 5 days
  * MDS patients >55 years receive 2.5 mg/kg/day for 5 days
  Other Names: ATG; Antithymocyte globulin
Drug: Cyclosporine — 5 mg/kg orally for 6 months; start after completing thymoglobulin.
  Other Names: CYA; Sandimmune; Cyclosporine A
Drug: Methylprednisolone — 1 mg/kg/day IV for 5 days, given before each dose of thymoglobulin.
  Other Names: Duralone®; Medralone®; Medrol®; M-Prednisol®; Solu-Medrol®
Drug: G-CSF — 5 microgram/kg subcutaneously daily up to 3 months, start after thymoglobulin.
  Other Names: Neupogen®; Granulocyte - Colony Stimulating Factor

SUMMARY:
The goal of this clinical research study is to learn if combining the drugs thymoglobulin, methylprednisolone, cyclosporine, and G-CSF (NeupogenTM or NeulastaTM ) can help to control severe aplastic anemia (AA) or hypoplastic myelodysplastic syndrome (MDS). The safety of this combination therapy will also be studied.

DETAILED DESCRIPTION:
Aplastic anemia is a condition that involves a low level of red blood cells (anemia), white blood cells, and platelets without evidence of another bone marrow disease. Anemia leads to fatigue, shortness of breath, and heart problems. Low platelet counts can lead to bruising and bleeding, and low white blood cell counts may cause an increased risk of infection, including pneumonia. Some of the treatment for AA includes transfusion, antibiotics and a combination of anti-thymocyte globulin (ATG) and cyclosporine with or without steroids, and growth factors such as G-CSF. For those who are eligible and have a donor, stem cell/bone marrow transplantation may be used.

MDS is a bone marrow disorder that usually affects older adults. Treatment of the bone marrow failure that accompanies MDS is usually with supportive care with red blood cell and platelet transfusions, antibiotics, and combinations of hematopoietic growth factors, which may partially improve blood cell counts.

It is often difficult to distinguish the hypoplastic variety of MDS from severe AA because both can result in bone marrow tests with very low cell count numbers. Earlier studies have shown that in some patients with the hypoplastic MDS, low blood counts respond to immunosuppressive treatment with ATG and cyclosporine. ATG is made from horse plasma. Thymoglobulin is a type of ATG made from rabbit plasma. Thymoglobulin has been successfully used to treat patients with AA who were previously treated with horse ATG but whose disease has returned. G-CSF is a growth factor that helps raise the white cell count after receiving chemotherapy. Methylprednisolone is a steroid that is commonly used in treating a number of medical conditions associated with people's abnormal immune response against themselves.

If you are found to be eligible to take part in this study, you will receive a combination of thymoglobulin, cyclosporine, G-CSF, and methylprednisolone. Treatment will be with thymoglobulin, which will be dosed depending on your age and weight. It will be given by vein over several hours once a day for a total of 5 days. You will receive the steroid methylprednisolone by vein before each dose of thymoglobulin to decrease the risk of developing allergic reactions to thymoglobulin. After 5 days of receiving methylprednisolone by vein, you will start taking it by mouth once a day at a decreasing dose over about 3 weeks.

The first 5 days of treatment will be given at M. D. Anderson but you will treated outside the hospital for the rest of the time unless complications develop.

You will be started on cyclosporine as well as G-CSF after completion of thymoglobulin. You will take cyclosporine by mouth twice a day for 6 months. Your physician may continue cyclosporine longer at his discretion. You will receive G-CSF as an injection under the skin for 3 months (or longer) once a day at the discretion of the treating physician starting at the same time as cyclosporine is started.

You will also receive antibiotic pills to help decrease the risk of infection. You will take levofloxacin, valacyclovir, fluconazole, or a similar antibiotic by mouth every day for the length of the study or until your treating physician finds appropriate.

If you have a history of heart disease and you take aspirin for this, your treating physician may consider stopping the aspirin because of your low platelet count as a result of your disease. This may increase your risk of heart attacks.

You will have blood tests (about 2 tablespoons each) once or twice a week for the first month and then once every 2-4 weeks until the end of the study to check if your blood counts are improving. The level of cyclosporine in your blood will also be checked at these times. It will require about 1 tablespoon for each of these tests. Monitoring of cyclosporine levels is a routine test done on all patients who receive this drug in order to avoid toxic blood levels and side effects.

At about 3 months, you will have a repeat bone marrow biopsy and aspiration as well as blood tests (about 3 tablespoons) to evaluate your response to the treatment.

You will continue cyclosporine for about 6 months (or longer if your doctor feels that it is in your interest) and will receive G-CSF for up to about 3 months (or longer if in your interest). If you develop serious side effects or if the disease gets worse at any time you will be taken off the study.

At the time when your doctor feels you have had the best possible response to the treatment and you are coming off study, blood tests (about 3 tablespoons) will be repeated.

Your doctor will continue to remain in touch with you to ensure that your disease remains under control. This may be done by arranging follow-up visits or through phone or other means of communication.

This is an investigational study. All the drugs used in this study are FDA approved and commercially available. Their use together in this study is experimental. A total of 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe aplastic anemia (bone marrow cellularity < 30%, with two of three peripheral counts at the time of initial presentation or currently low with absolute neutrophil count (ANC) < 500/mL, pre-transfusion platelet (PLT) < 20,000/mL, or pre-transfusion hemoglobin < 8 g/dL and presence of no other underlying disorder.
* Diagnosis of MDS (World Health Organization) with bone marrow cellularity < 30%, with two of three peripheral counts at the time of initial presentation or currently low with ANC < 500/mL, pre-transfusion PLT < 20,000/mL, or pre-transfusion hemoglobin < 8 g/dL.
* Patients with MDS who have received prior biological therapy (not chemotherapy) are eligible. Hypomethylating agents and histone deacetylase inhibitors are considered as biological therapy.
* Age 15 or greater
* Adequate renal function (creatinine less than or equal to 2.0 mg/dL) unless related to the disease
* Adequate hepatic function (bilirubin less than or equal to 3.5 mg/dL) unless related to the disease
* No other investigational therapy in the past 14 days
* Able to sign consent form
* Able to comply with the need for contraception (abstinence, condom, birth control pill, or other acceptable form of contraception) during the entire study period
* Diagnosis of MDS (WHO) with bone marrow cellularity greater than 30%, with low or intermediate-1 risk by the International Prognostic Scoring System (IPSS) score, and requiring treatment (i.e. transfusion-dependent)

Exclusion Criteria:

* Active and uncontrolled infection
* HIV positive test
* Pregnant or breast feeding
* Active and uncontrolled medical illness (pulmonary, cardiac, neurological, or other) that in the opinion of treating physician would likely interfere with study treatment

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tapan M. Kadia, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 5/12/2005 - 6/20/2012; all participants were registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: A total of 53 participants were enrolled on the study, with four patients choosing alternative treatment; one participant died before administration of study treatment.
Groups:
- Thymoglobulin + Cyclosporin: Combination of Thymoglobulin + Methylprednisone + Cyclosporin + G-CSF
  Cyclosporine : 5 mg/kg orally for 6 months; start after completing thymoglobulin.
  G-CSF : G-CSF 5 microgram/kg subcutaneously daily up to 3 months, start after thymoglobulin.
  Thymoglobulin : 3.5 or 2.5 mg/kg/day IV for 5 days
  * Aplastic anemia patients receive 3.5 mg/kg/day for 5 days
  * MDS patients <55 years receive 3.5 mg/kg/day for 5 days
  * MDS patients >55 years receive 2.5 mg/kg/day for 5 days
  Methylprednisolone : 1 mg/kg/day IV for 5 days, given before each dose of thymoglobulin.
Period: Overall Study
Arm/Group | Thymoglobulin + Cyclosporin
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Thymoglobulin + Cyclosporin
Number analyzed (Participants) | 48
Age Continuous [Median (Full Range); unit: years] | 59 [19 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Complete response (CR) was defined as normalization of peripheral blood and bone marrow with <5% blasts, a peripheral absolute neutrophil count (ANC) >/= 1 * 10^9/l, hemoglobin >/= 100g/l, and a platelet count >/= * 10^9/l, Partial Response (PR) was defined as transfusion independence with a peripheral blood ANC >=/ 0.05 * 10^9/l, a platelet count >/= 20 * 10^9/l, and a hemoglobin >/= 40 g/l. Hematologic improvement was defined as a clinically relevant increase in hemoglobin, platelets or absolute neutrophil count.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first. Assessed first at 3 months on study, continuing monthly up to 3 years.
Population: Of the 48 participants who received treatment 46 were evaluable for response.
Measure: Number; unit: participants
Groups:
- Thymoglobulin + Cyclosporin: Combination of Thymoglobulin + Methylprednisone + Cyclosporin + Granulocyte Colony stimulating factor (G-CSF
  Cyclosporine : 5 mg/kg orally for 6 months; start after completing thymoglobulin.
  G-CSF : G-CSF 5 microgram/kg subcutaneously daily up to 3 months, start after thymoglobulin.
  Thymoglobulin : 3.5 or 2.5 mg/kg/day IV for 5 days
  * Aplastic anemia patients receive 3.5 mg/kg/day for 5 days
  * MDS patients <55 years receive 3.5 mg/kg/day for 5 days
  * MDS patients >55 years receive 2.5 mg/kg/day for 5 days
  Methylprednisolone : 1 mg/kg/day IV for 5 days, given before each dose of thymoglobulin.
Arm/Group | Thymoglobulin + Cyclosporin
Number analyzed (Participants) | 46
participants
  Complete Response | 8
  Partial Response | 8
  Hematological Improvement | 4

ADVERSE EVENTS:
Time Frame: Seven years, one month
Arm/Group | Thymoglobulin + Cyclosporin
Serious Adverse Events (participants affected / at risk) | 8/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thymoglobulin + Cyclosporin (N=48)
Fever (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Infection (Infections and infestations) | 3 (3)
Neutropenic Fever (Infections and infestations) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Death (General disorders) | 2 (2)
Prolonged Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Respiratory Alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal Pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thymoglobulin + Cyclosporin (N=48)
Neutropenia (Blood and lymphatic system disorders) | 24 (24)
Thrombocytopenia (Blood and lymphatic system disorders) | 22 (22)
Elevated Creatinine (Renal and urinary disorders) | 19 (19)
Elevated Transaminases (Hepatobiliary disorders) | 16 (16)
Elevated Bilirubin (Hepatobiliary disorders) | 15 (15)
Anemia (Blood and lymphatic system disorders) | 13 (13)
Elevated Uric Acid (Metabolism and nutrition disorders) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 7 (7)
Fatigue (General disorders) | 6 (6)
Low Magnesium (Metabolism and nutrition disorders) | 6 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Nausea/Vomining (Gastrointestinal disorders) | 5 (5)
Low Potassium (Metabolism and nutrition disorders) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5)
Low Sodium (Metabolism and nutrition disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Edema (General disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Infusion Reaction (General disorders) | 23 (23)
Infection (Infections and infestations) | 10 (10)
Neutropenic Fever (Infections and infestations) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes